CLINICAL TRIAL: NCT03616262
Title: "Efficacy of Botulinum Toxin Injection in Reducing Limb Pain in Patients With Complex Regional Pain Syndrome"
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VACHS
Record Dates: First submitted 2015-07-13; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-07

CONDITIONS: Complex Regional Pain Syndrome
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Botulinum Toxins, Type A; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Active Comparator): In Phase 1, subjects will receive either Treatment A (Lidocaine alone) or Treatment B (Botox+Lidocaine )
  Interventions: Drug: Botox + Lidocaine; Drug: Lidocaine alone
- Phase 2 (Active Comparator): In Phase 2, subjects will receive either Treatment B (Botox+Lidocaine) or Treatment A (Lidocaine alone) -- the opposite of what was administered in Phase 1
  Interventions: Drug: Botox + Lidocaine; Drug: Lidocaine alone

INTERVENTIONS:
Drug: Botox + Lidocaine — The total dose per patient in the lower extremity or upper extremity will be based on common doses given in spasticity patients in the neurology injection clinic. If the target is a symptomatic arm, we will inject as follows: biceps 30 units, triceps 40 units, flexor carpi radialis 20 units, extensor carpi radialis 20 units. If the target is a symptomatic leg, we will inject in the following pattern: vastus lateralis 50 units, rectus femoris 30 units, medial gastrocnemius 40 units, tibialis anterior 40 units.
Drug: Lidocaine alone — The total dose per patient in the lower extremity or upper extremity will be based on common doses given in spasticity patients in the neurology injection clinic. If the target is a symptomatic arm, we will inject as follows: biceps 30 units, triceps 40 units, flexor carpi radialis 20 units, extensor carpi radialis 20 units. If the target is a symptomatic leg, we will inject in the following pattern: vastus lateralis 50 units, rectus femoris 30 units, medial gastrocnemius 40 units, tibialis anterior 40 units.

SUMMARY:
Objective: The primary aim is to evaluate the efficacy of botulinum toxin A in reducing overall limb pain in patients with complex regional pain syndrome (CRPS). Additionally the investigators would like to see if quality of life is improved and disability scores decreased.

Research Design:

This is a double blinded, randomized cross-over study that will be conducted over a 7 month period. It is a pilot study that will include twenty subjects recruited from the Neurology CRPS clinic at VA Connecticut and from outside VA hospitals within a 150 mile radius. Subjects will receive an intramuscular injection Treatment A which is only 1% lidocaine or Treatment B which is mixture of botulinum toxin A + 1% lidocaine in the affected limb only. This is a cross over study where patients will receive Treatment A or B initially during the first of four study visits and during the third study visit while receive whichever treatment not given during the first visit. Dr. Sameer Ali, VA neurology fellow, will be blinded when administering the treatments. Dr. Hajime Tokuno, VA neurologist who is the principal investigator of the trial will prepare the treatments. Clinical pharmacy will be randomizing the treatments. Dr. Tokuno will not be blinded as he needs to know which treatment has been given in case of complications.

Impact/Significance: The significance of this study is the possible discovery of a new, safer, less invasive, and more efficacious therapeutic option for patients suffering from CRPS. Currently medical management with neuropathic pain meds, interventions such as sympathetic nerve blocks and ketamine infusion has helped some patients and not others. The investigators are trying to see whether either of the two treatments and especially the treatment with botulinum toxin may be a more viable alternative than existing modalities.

DETAILED DESCRIPTION:
PROJECT DESCRIPTION Principal Investigator: Hajime Tokuno, MD

Project Title: "Efficacy of botulinum toxin injection in reducing limb pain in patients with Complex Regional Pain Syndrome"

Purpose: Complex Regional Pain Syndrome is a condition affecting anywhere from 1 to 5 million Americans including members of our veteran population for which there are woefully few effective therapeutics options. The investigators hypothesize that they can reduce overall pain levels in patients with Complex Regional Pain Syndrome (CRPS) using botulinum toxins. Reduction in the VAS score will be the primary outcome measure. Additionally they hypothesize that the quality of life will improve and disability will decrease, thus these two parameters both quality of life and disability will serve as the main secondary outcome measures. Additional secondary outcome measures include thermography, goniometry, algometry, electrical impedance myography, and a modified VAS scale designed by the investigators.

Background:

CRPS is a poorly defined medical entity that consists of a number of different signs and symptoms including neuropathic pain (or allodynia), ischemic pain, sympathetically mediated pain, and myofascial pain. There have been a number of therapeutic options such as anticonvulsants to treat neuropathic pain. Sympathetic mediated central pain has been treated with sympathetic ganglion blocks.

There are two similar forms called CRPS-I and CRPS-II with the same symptoms and treatments. CRPS-I has previously been known as RSD or Reflex Sympathic Dystrophy Syndrome and involves individuals without confirmed nerve injury. CRPS-II has previously been known as causalgia and involves individuals whose symptoms appeared after a confirmed nerve injury.

CRPS can appear at any age. It is rare in the elderly and more common in women. Occasionally CRPS can develop without any known injury. There is no specific single diagnostic test to confirm CRPS and diagnosis is made based on the affected individual's medical history and signs/symptoms that match the definition; it is a diagnosis of exclusion. (Borchers 2014).

The component of CRPS largely ignored has been the myofascial pain component. Patients in the VA CRPS clinic at West Haven, CT have been found to have a myofascial pain component and responded positively to Botox injections. In one anecdotal case, the patient claimed that botulinum toxin injection was the only drug that ever helped her overall pain albeit in a limited fashion. Botulinum toxins are compounds known to relax tightly contracted muscles by blocking the release of acetylcholine, the sole neurotransmitter that initiates muscle contraction at the neuromuscular junction (Kalandakanond & Coffield 2001). They are a well-established class of neurotoxin with a wide variety of FDA approved medical applications including muscle relaxation, headache prevention and bladder control (Chen 2012). There are only a handful of studies assessing botulinum toxin A injections for the treatment of CPRS related pain. The results are mixed. There are two studies utilizing intramuscular botulinum toxin, one by Safarpour et al 2010 comprising of two patients and the other by Argoff 2002 consisting of 11 patients. Patients demonstrated overall pain improvement with the intramuscular Botox injections similar to the investigators' results.

In this study, the investigators are utilizing four novel devices; goniometry to assess range of motion of the upper or lower extremity limb joints, infrared thermography to assess heat production in affected body regions, algometry to quantify pressure-pain thresholds, and electrical impedance myography to assess atrophy in a quantitative manner.

A goniometer is a simple mechanical tool used by physiotherapists that can quickly and safely assess passive range of motion of individual limb joints. The units of measure will be recorded in degrees change from the resting position to the fully flexed or extended position for a given joint. For upper extremity CPRS, the investigators will assess arm flexion, arm extension, wrist extension, wrist flexion for both the affected limb as well as the normal limb. The normal will serve as the internal control. For lower extremity CRPS, they will assess leg flexion, leg extension, dorsiflexion, plantar flexion. They will obtain a measure of rotational range of motion of a joint using degrees of change compared to the unaffected limb.

The investigators will be using a digital goniometer known as the Baseline Absolute Axis 360 Degree Goniometer. For this study, one physical therapist will carry out all the measurements in order to avoid inter-examiner variability. She will obtain the mean of 3 separate measurements at each joint.

Digital infrared thermography can record heat emanation from pre-defined regions of interest (ROI) in affected area of the body, non-invasively. Studies of CRPS suggest that limb temperatures are often elevated acutely and decreased chronically. There are mixed results regarding the utility of thermography in the diagnosis of CRPS and the investigators of this study are hoping to provide further insight into this matter. Because of the mixed results of infrared imaging in pain patients (Ra et al 2013), they will use this parameter as a secondary outcome measure. The specific device they will be utilizing is a FLIR A65 series medical grade IR thermography unit. They will be utilizing quantitative thermography where they will utilize the selected regions of interest (ROIs) and compare between the affected and unaffected areas on the contralateral limb(s). They will be utilizing the Research IR Max software to perform statistical analyses. Below are the defined ROIs:

flexor carpi radialis and flexor digitorum superficialis, extensor carpi radialis and extensor carpi ulnaris, biceps, triceps, anterior compartment leg muscles, gastrocnemii quadriceps hamstrings and hip adductors.

They have developed these ROIs based on their own observations in the CRPS clinic. They have observed that the limb hypothermia localizes mostly to the large proximal muscles on the side of a hand or foot experiencing allodynia. There was less correlation with the affected distal limb segment where the allodynia was perceived. Similar observations were made by a group that examined the reliability of IRT in the diagnosing CRPS (Choi et al 2013).

An algometer is a device that measures pain thresholds in affected areas. The investigators will be utilizing a digital algometer designed by Wagner Instruments called the Force One Digital Force Gauge. They will be recording the minimal pressure required to trigger a pain response at several pre-designated site. The physical therapist on their team will obtain the measurements and will record the average of three readings. The operator of the device will apply a steady force at a predefined site on an affected limb, and a digital readout of the pain threshold will be recorded in kilopascal units (kPa = Newtons/m2) per second. They will utilize the same muscle groups laid out in the ROIs above. In all instances, the central belly of the muscle will be targeted and pressure will be applied to the central belly until the patient perceives pain at that site. The pressure readout will be recorded for later comparison and correlation with other primary and secondary measures. They are focusing on the central belly because this is where the majority of trigger points are located (Margoles 1999).

They will also utilize electrical impedance myography (EIM) in this study. EIM assesses disease-induced changes in muscle tissue, including myocyte atrophy and loss, muscle edema, and fatty infiltration. It is a new technology that is non invasive and safe. EIM uses high-frequency, low intensity electrical currents to quantify disuse atrophy and other muscle pathology. The low intensity of the current prevents the muscle and nerve depolarization threshold, and therefore, the patient experiences no unpleasant sensation during the study. This is especially important with the CRPS patients who are chronically experiencing tremendous pain. Rutkove et al demonstrated that leg atrophy following limb immobilization as well as restoration of normal muscle bulk was measureable with an EIM device. Rutkove used a parameter was called θ which is a measure of both resistance and capacitance θ = arctan (X/R) where X = 1/capacitance and R = resistance.

The investigators wish to quantify the muscle atrophy in CRPS patients using the same technology. Clinical experience has shown that the painful limbs are often atrophic and cold. The investigators are interested in understanding the relationship between heat production and muscular atrophy and if EIM can give them a more precise and representation of this phenomenon. (Tarulli et al 2009).

Significance:

The potential benefits are overall pain reduction in the painful extremity as demonstrated by reduced score on the VAS. Additionally there may be improvement of quality of life and reduction in disability. This project may contribute to the utilization of a new treatment modality for CRPS that may reduce limb pain more so than any current modality.

Research Plan:

Methods:

This is a double blinded, randomized cross-over study that will be conducted over an estimated 7 month period for each study participant. It is a pilot study that will include twenty subjects recruited from the Neurology CRPS clinic at VA Connecticut and also from the area VA hospitals within a 150 mile radius. Subjects will receive an intramuscular injection Treatment A which is only 1% lidocaine or Treatment B which is mixture of botulinum toxin A + 1% lidocaine in the affected limb only. This is a cross over study where patients will receive Treatment A or B initially during the first of four study visits and during the third study visit will receive whichever treatment not given during the first visit. Dr. Sameer Ali, VA neurology fellow, will be blinded when administering the treatments. Dr. Hajime Tokuno, VA neurologist who is the principal investigator of the trial will prepare the treatments. Clinical pharmacy will be randomizing the treatments. Dr. Tokuno will not be blinded as he needs to know which treatment has been given in case of complications.

The total dose of Treatment A or B per patient in the lower extremity or upper extremity will be based on common doses given in spasticity patients in the neurology injection clinic. The total dose per patient in the arm will be as follows: biceps 30 units, triceps 40 units, flexor carpi radialis 20 units, extensor carpi radialis 20 units. The total dose per patient in the leg will be as follows: vastus lateralis 50 units, rectus femoris 30 units, medial gastrocnemius 40 units, tibialis anterior 40 units. The dosing pattern will be largely exam dependent as we will inject the actual areas or proximal to the areas that are painful either at rest or upon stretch. A maximum of 200 units of botulinum toxin A will be administered at a time as to minimize the risk of side effects.

For the treatment B arm one vial of ONABOTULINUMTOXINA 200 UNITS/VIAL for each subject will be drawn in two separate syringes of 100 units each and reconstituted with the 1% lidocaine. For treatment A there will be two syringes filled with 1% lidocaine. Dr. Tokuno will prepare the treatments and randomization and storage will be provided by the clinical pharmacy. The reconstituting will be done in the clinic. Patients will be injected at the VA Connecticut during CRPS clinic hours.

There will be a washout period of 4 months for the patients receiving the first round of injections (lidocaine or botulinum toxin + lidocaine) prior to the crossover. There will be a total of 4 visits to the VA. The first visit-either injection of Treatment A or B, the post injection 1 month follow up. After 3 more months have gone by (4 months post injection=washout period) then the treatment arm will switch and pt will again come in for the injection and post injection 1 month follow up.

All four study visits will start with obtaining the VAS score, a modified VAS score we have designed, pain disability index and quality of life scores. We will utilize a modified VAS scale to ask patient the average level of pain in a day, the lowest and highest pain scores for that day, and the exact contributions of various qualities of the pain specifically myofascial and hypersensitivity pain.

We then will proceed by obtaining data with the utilization of thermography, goniometry, algometry, EIM. Thermographic data will allow us to look at heat production in the affected limb compared to unaffected limb and if there is a change after treatment A or B when reassessed. Algometry will allow us to determine how much pressure is needed to allow for realization of discomfort and if this changes post treatment. Goniometry will allow us to determine the range of motion of both affected and unaffected muscles to see if there is a difference as we are expecting decreased range in the affected limb. We can then see if the range of motion will improve after either treatment. We also will utilize EIM to assess if our treatments can alter changes of impedance in the affected limb.

The primary outcome measure is pain reduction reflected by the VAS scale and the secondary outcome measures are quality of life and disability as well as thermography and range of motion. This study will test the effects of a one-time botulinum toxin A injection.

Statistical analysis-. We will have patients come one month after each of the two injections to reassess their functional status using goniometry, thermography and neurologic exam. The primary outcome measure is pain reduction reflected by the VAS scale and the secondary outcome measures are quality of life and disability as well as thermography and range of motion. This study will test the effects of a one-time botulinum toxin A injection. The Pierson product-moment correlation will be used to assess the pain via the VAS score over time. The Spearman rank-order correlation will be used to assess the VAS scale and the following secondary outcome measures-Range of motion, thermography, quality of life, disability.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with documented diagnosis of CRPS per International Pain Society Guidelines. Diagnosis must be made or confirmed in the neurology CRPS clinic prior to recruitment.
2. Patients ages 18-80.
3. Patients may or may not have tried other therapeutics, will not affect study.
4. Veterans enrolled in the Veterans Hospital system of the United States.
5. Patients enrolled either type I or II CRPS of either upper or lower extremity.

Exclusion Criteria:

1. Prior history of adverse side effects with use of botulinum toxin.
2. Prior adverse reaction to lidocaine use.
3. CRPS involving multiple extremities.
4. Myasthenia gravis, myopathy, severe polyneuropathy or other causes of chronic muscle weakness.
5. History of severe mental illness or dementia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in the VAS score will be the primary outcome measure. | 7 months
  The VAS score will be obtained using the VAS at each of the four study visits. Zero is no pain and ten is maximum pain on the zero to ten scale.

SECONDARY OUTCOMES:
Quality of Life as a measure of function with pain. | 7 months
  The Quality of Life scale will be utilized at each of the four study visits. We will be paying attention to change in the quality of life during this study. This scale is a measure of function for people with pain. zero=non functioning, ten=normal quality of life.
Disability | 7 months
  The Pain Disability Index scale will be utilized at each of the four study visits. We will be paying attention to change in disability during this study. This scale is designed to measure the degree that seven aspects of life are disrupted by chronic pain. These seven aspects are family/home responsibilities, recreation, social activity, occupation, sexual behavior, self care, life-support activities. This is a zero to ten scale with zero=no disability, and ten=worst disability.
Thermography | 7 months
  Digital infrared thermography can record heat emanation from pre-defined regions of interest (ROI) in affected area of the body, non-invasively. . The specific device that we will be utilizing is a FLIR A65 series medical grade IR thermography unit.
Goniometry | 7 months
  A goniometer (a.k.a. inclinometer) is a simple mechanical tool used by physiotherapists that can quickly and safely assess passive range of motion of individual limb joints. Contracture or dystonia of associated muscles will reduced the range of motion of the joint. The units of measure will be recorded in degrees change from the resting position to the fully flexed or extended position for a given joint. We will be using a digital goniometer known as the Baseline Absolute Axis 360 Degree Goniometer.
Algometry | 7 months
  An algometer is a device that measures pain thresholds in affected areas. We are recording the minimal pressure required to trigger a pain response at several pre-designated sites. The operator of the device will apply a steady force at a predefined site on an affected limb, and a digital readout of the pain threshold will be recorded in kilopascal units (kPa = Newtons/m2) per second. We will be utilizing a digital algometer designed by Wagner Instruments called the Force One Digital Force Gauge.
Modified VAS Score | 7 months
  This has been designed by our research team. This is comprised of asking for the average level of pain, lowest level of pain, highest level of pain for the day, allodynia, muscular pain component. These components are based on zero being no pain and ten being maximum pain on the zero to ten scale.
Electrical Impedence Myography | 7 months
  EIM assesses disease-induced changes in muscle tissue, including myocyte atrophy and loss, muscle edema, and fatty infiltration. It is new technology that is non invasive and safe. EIM uses high-frequency, low intensity electrical currents to quantify disuse atrophy and other muscle pathology.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

REFERENCES:
- [Background] Argoff CE. A focused review on the use of botulinum toxins for neuropathic pain. Clin J Pain. 2002 Nov-Dec;18(6 Suppl):S177-81. doi: 10.1097/00002508-200211001-00010. PMID 12569966
- [Background] Birthi P, Sloan P, Salles S. Subcutaneous botulinum toxin A for the treatment of refractory complex regional pain syndrome. PM R. 2012 Jun;4(6):446-9. doi: 10.1016/j.pmrj.2011.12.010. No abstract available. PMID 22732156
- [Background] Borchers AT, Gershwin ME. Complex regional pain syndrome: a comprehensive and critical review. Autoimmun Rev. 2014 Mar;13(3):242-65. doi: 10.1016/j.autrev.2013.10.006. Epub 2013 Oct 23. PMID 24161450
- [Background] Choi E, Lee PB, Nahm FS. Interexaminer reliability of infrared thermography for the diagnosis of complex regional pain syndrome. Skin Res Technol. 2013 May;19(2):189-93. doi: 10.1111/srt.12032. Epub 2013 Jan 20. PMID 23331254
- [Background] Chen S. Clinical uses of botulinum neurotoxins: current indications, limitations and future developments. Toxins (Basel). 2012 Oct;4(10):913-39. doi: 10.3390/toxins4100913. Epub 2012 Oct 19. PMID 23162705
- [Background] Jeong MY, Yu JS, Chung WB. Usefulness of thermography in diagnosis of complex regional pain syndrome type I after transradial coronary intervention. J Invasive Cardiol. 2013 Sep;25(9):E183-5. PMID 23995728
- [Background] Kalandakanond S, Coffield JA. Cleavage of SNAP-25 by botulinum toxin type A requires receptor-mediated endocytosis, pH-dependent translocation, and zinc. J Pharmacol Exp Ther. 2001 Mar;296(3):980-6. PMID 11181932
- [Background] Niehof SP, Huygen FJ, Stronks DL, Klein J, Zijlstra FJ. Reliability of observer assessment of thermographic images in complex regional pain syndrome type 1. Acta Orthop Belg. 2007 Feb;73(1):31-7. PMID 17441655
- [Background] Niehof SP, Beerthuizen A, Huygen FJ, Zijlstra FJ. Using skin surface temperature to differentiate between complex regional pain syndrome type 1 patients after a fracture and control patients with various complaints after a fracture. Anesth Analg. 2008 Jan;106(1):270-7, table of contents. doi: 10.1213/01.ane.0000289635.95869.70. PMID 18165590
- [Background] Ra JY, An S, Lee GH, Kim TU, Lee SJ, Hyun JK. Skin temperature changes in patients with unilateral lumbosacral radiculopathy. Ann Rehabil Med. 2013 Jun;37(3):355-63. doi: 10.5535/arm.2013.37.3.355. Epub 2013 Jun 30. PMID 23869333
- [Background] Safarpour D, Jabbari B. Botulinum toxin A (Botox) for treatment of proximal myofascial pain in complex regional pain syndrome: two cases. Pain Med. 2010 Sep;11(9):1415-8. doi: 10.1111/j.1526-4637.2010.00929.x. Epub 2010 Aug 23. PMID 20735753
- [Background] Safarpour D, Salardini A, Richardson D, Jabbari B. Botulinum toxin A for treatment of allodynia of complex regional pain syndrome: a pilot study. Pain Med. 2010 Sep;11(9):1411-4. doi: 10.1111/j.1526-4637.2010.00897.x. Epub 2010 Jun 30. PMID 20609130
- [Background] Shahidi B, Johnson CL, Curran-Everett D, Maluf KS. Reliability and group differences in quantitative cervicothoracic measures among individuals with and without chronic neck pain. BMC Musculoskelet Disord. 2012 Oct 31;13:215. doi: 10.1186/1471-2474-13-215. PMID 23114092